CLINICAL TRIAL: NCT00447109
Title: Endotracheal Suction With or Without Daily Changes of Closed System Suction. Effect on Ventilator Associated Pneumonia and Cost
Brief Title: Time Interval for Changing Closed System Suction Catheters, Effect on Ventilator Associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Deakin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122/02; T10308
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2007-03-14 (Estimated); Status verified 2007-03

CONDITIONS: Pneumonia, Ventilator Associated; Closed System Suction Catheter
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Closed system suction

SUMMARY:
The purpose of this study was to compare the incidence of ventilator-associated pneumonia between two groups of patients randomised to have closed system suction catheter changes every 24 hours and patients having closed system suction catheter changes every seven days or as required.

DETAILED DESCRIPTION:
Comparison(s): the incidence of ventilator-associated pneumonia between two groups of patients randomised to have closed system suction catheter changes every 24 hours and patients having closed system suction catheter changes every seven days or as required.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than 18 years
* Mechanically ventilated for more than 24 hours

Exclusion Criteria:

* Admitted from other hospital already mechanically ventilated
* Massive haemoptysis
* Previously received mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 344
Dates: Start 2003-09; Study Completion 2004-04

PRIMARY OUTCOMES:
ventilator-associated pneumonia

SECONDARY OUTCOMES:
length of hospital
intensive care stay
duration of mechanical ventilation
hospital mortality
number of acquired organ system derangements
cost of the closed system suction catheters

CONTACTS AND LOCATIONS:
Overall Officials: Lauren J McTier, Principal Investigator — Deakin University
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia